CLINICAL TRIAL: NCT05259800
Title: Evaluating the Use of Peppermint Oil for Postpartum Women With Urinary Retention
Brief Title: Peppermint Oil for Urinary Retention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty enrolling patients
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-065
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Urinary Retention
Keywords: peppermint oil; postpartum
MeSH Terms: conditions — Urinary Retention | interventions — Mineral Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peppermint Oil (Experimental): Subjects will be exposed to vapor of peppermint oil
  Interventions: Other: Peppermint oil vapors
- Placebo (Placebo Comparator): Subjects will be exposed to vapor of placebo (mineral oil)
  Interventions: Other: Mineral Oil

INTERVENTIONS:
Other: Peppermint oil vapors — Subjects will be exposed to vapor of peppermint oil
  Arms: Peppermint Oil
Other: Mineral Oil — Subjects will be exposed to vapor of placebo (mineral oil)
  Arms: Placebo

SUMMARY:
A randomized controlled study will be conducted, with two arms. Postpartum women experiencing urinary retention will be randomized into one of the two following arms:

* Arm 1: Subjects will be exposed to vapor of peppermint oil
* Arm 2: Subjects will be exposed to vapor of placebo (mineral oil) Outcome variables include resolution of urinary retention, time to spontaneous urination, volume of spontaneous urination, frequency of urinary catheterization, and patient satisfaction.

DETAILED DESCRIPTION:
The purpose of the study is to determine if the use of peppermint oil among postpartum women experiencing urinary retention will increase spontaneous urination and decrease the need for catheterization. A randomized controlled study will be conducted, with two arms. Subjects will be randomized into one of the two following arms:

* Arm 1: Subjects will be exposed to vapor of peppermint oil
* Arm 2: Subjects will be exposed to vapor of placebo (mineral oil) Outcome variables include resolution of urinary retention, time to spontaneous urination, volume of spontaneous urination, frequency of urinary catheterization, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 years old or older 2. English speaking 3. Admitted to Bethesda North Mom Baby Unit 4. Postpartum 5. Experiencing urinary retention - defined as meeting at least one of the following criteria:

  * More than 6 hours after delivery or foley catheter removal without being able to spontaneously void
  * Symptomatic urinary retention without being able to spontaneously void
  * Change in fundal height or position without being able to spontaneously void 6. Bladder scan showing bladder containing 400mL or more urine

Exclusion Criteria:

1. Allergy to peppermint
2. Asthma
3. Active herpes lesions
4. Seizure disorder
5. Not able to void in toilet (ex: requiring use of bed pan to void)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Postpartum women
Enrollment: 17 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bethesda North Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peppermint Oil | Placebo
Started | 10 | 7
Completed | 10 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peppermint Oil | Placebo | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 7 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With Urinary Retention Resolved
Description: Urinary retention defined as:
  * More than 6 hours after delivery or foley catheter removal without being able to spontaneously void
  * Symptomatic urinary retention without being able to spontaneously void
  * Change in fundal height or position without being able to spontaneously void More than 6 hours after delivery or foley catheter removal without voiding spontaneously; symptomatic urinary retention without being able to spontaneously void; or change in fundal height or position without being able to spontaneously void
  Resolution of urinary retention will be achieved if patient spontaneously voids within 10 minutes after exposure to oil
Time Frame: 10 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Peppermint Oil | Placebo
Number analyzed (Participants) | 10 | 7
Participants | 3 | 1

2. Secondary Outcome: Time to Spontaneous Urination
Description: Minutes until participant spontaneously voids
Time Frame: 1 hour
Reporting Status: Not Posted

3. Secondary Outcome: Volume of Spontaneous Urination
Description: Volume of urine when participant spontaneously voids
Time Frame: 1 hour
Reporting Status: Not Posted

4. Secondary Outcome: Incidence of Urinary Catheterization
Description: Whether participant requires urinary catheterization or not
Time Frame: 1 hour
Reporting Status: Not Posted

5. Secondary Outcome: Patient Satisfaction
Description: Patient rated satisfaction
Time Frame: 1 hour
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, up to 2 days
Arm/Group | Peppermint Oil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 0/10 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT05259800/Prot_SAP_000.pdf